CLINICAL TRIAL: NCT00104455
Title: Recombinant Activated Factor VII (rFVIIa/NovoSeven) Dose Response Trial in Healthy Volunteers: A Double-Blind, Placebo-Controlled, Cross-over, Dose-Escalation Trial to Investigate the Dose Response to REcombinant Factor VIIa When Administered for Bleeding Following Punch Biopsies in Healthy Volunteers
Brief Title: Dose Response to Recombinant Factor VIIa When Administered for Bleed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7DRC-2157
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Healthy
Keywords: rFVIIa; Punch Biopsy; Dose Response; Healthy People Programs

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of this trial is to investigate the dose response to recombinant factor VIIa in healthy volunteers when administered for bleed.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years - 60 Years

Exclusion Criteria:

* - -

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2004-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Dose Response to Recombinant Factor VIIa

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Result] Gabriel DA, SKolnick BE, S Seremitis, Leese P, Mathews D. Effect of Recombinant Activated Factor VII (rFVIIa) on Platelet and Clotting Systems in Healthy Volunteers. Blood 2005; 106 (11): Abstract No. 4053
- [Result] Gabriel DA, Skolnick BE, Rojkjaer LP, Seremetis SV. Variations in Ex-Vivo Assessments of Hemostasis. Blood 2005; 106 (11): Abstract No. 4052
- [Result] Gabriel DA, Skolnick BE, Leese P, Mathews D. Ex-vivo Assessments in the Evaluation of Dose Response to Recombinant Factor VIIa when Administered for Bleeding Following Punch Biopsies in Healthy Volunteers. Blood 2005; 106 (11): Abstract No. 4055
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com